CLINICAL TRIAL: NCT01654445
Title: A Phase 2, Prospective, Two Cohort, Dose-escalation, Safety and Feasibility Study of Thrombolysis for Minor Ischemic Stroke With Proven Acute Symptomatic Occlusion Using TNK-tPA
Brief Title: TNK-tPA Evaluation for Minor Ischemic Stroke With Proven Occlusion
Acronym: TEMPO-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Vancouver General Hospital (Other); Ottawa Hospital Research Institute (Other); Hopital Charles Lemoyne (Other); Université de Sherbrooke (Other); Vancouver Island Health Authority (Other); CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Dr. Michael Hill, PI, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Version 2.2, Aug 28,2013
Record Dates: First submitted 2012-07-25; First posted 2012-07-31 (Estimated); Results first posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Ischemic Stroke
Keywords: Minor stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Tenecteplase; TNK-tissue plasminogen activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TNK-tPA Tenecteplase (Experimental): This is an open-label trial, all patients will receive tenecteplase.
  Interventions: Drug: Tenecteplase

INTERVENTIONS:
Drug: Tenecteplase — Tenecteplase will be given to the patient as an intravenous bolus over 1- 2 minutes within 90 minutes of the first slice of the CTA. This is an open-label trial, all patients will receive tenecteplase, either tier 1 or tier 2 dosage.
  Other Names: TNK-tPA

SUMMARY:
This trial will enroll patients that have been diagnosed with a transient ischemic attack (TIA) or minor stroke that has occurred within the past 12 hours. Anyone diagnosed with a minor stroke faces the possibility of long-term disability and even death, regardless of treatment. Stroke symptoms such as weakness, difficulty speaking and paralysis may improve or worsen over the hours or days immediately following a stroke. The purpose of this research trial is to study the effects of a clot-dissolving drug, tenecteplase (TNK-tPA), as a treatment for patients who arrive within twelve hours from stroke onset. This study is attempting to see if TNK-tPA given through a vein in the arm (intravenous) to patients is a safe treatment for stroke patients. Neither the safety nor the effectiveness of this treatment has been proven yet.

This trial will be conducted at several site in Canada.

Dr Michael Hill and Dr. Shelagh Coutts are the Principal Investigators of this trial, coordinated at the University of Calgary, Foothills Medical Centre.

DETAILED DESCRIPTION:
The primary objective of TEMPO-1 is to demonstrate the safety and feasibility of using TNK-tPA (tenecteplase), a thrombolytic agent that is relatively novel to the treatment ischemic stroke but well-established in the treatment of myocardial infarction, to treat minor ischemic stroke patients with proven acute symptomatic occlusions. Up to 80% of ischemic stroke is minor and initially non-disabling. These patients present with a transient ischemic attack (TIA) or minor stroke.An overwhelming majority are not treated with thrombolysis as they are considered "too good to treat" by most physicians.

TEMPO-1 will enroll patients within a 12 hour time window with a NIHSS score of <6 and an ASPECTS >5. Patients must have an intracranial occlusion on CTA. Study drug must be administered within 90 minutes from the first slice of CTA. This is an open- label, multi-centre trial, dose- escalated trial. A total of 50 patients will be enrolled, 25 per tier. There will two dose tiers at 0.1 mg/kg and 0.25 mg/kg. Advancement to the second dose-tier will be dependent upon safe completion of the 1st dose tier and the approval of the DSMB.

Patients will undergo a study CT angiogram of the intracranial circulation between 4-8 hours after treatment to determine the biological effect of the drug - whether the occluded artery has recanalized or not. Patients will be assessed at 24 and 48 hours, and at Days 5, 30, and 90.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke in an adult patient (18 years of age or older)
2. Onset (last-seen-well) time to treatment time < 12 hours.
3. Minor stroke defined as a baseline NIHSS < 6 at the time of randomization. Patients must have a demonstrable neurological deficit on physical neurological examination.
4. Any acute intracranial occlusion (MCA, ACA, PCA, VB territories) defined by non-invasive acute imaging (CT angiography) that is neurologically relevant to the presenting symptoms and signs. An acute occlusion is defined as TICI 0 or TICI 1 flow.
5. Pre-stroke independent functional status in activities of daily living with pre-stroke estimated modified Barthel Index of 90 or greater AND premorbid mRS 0 or 1.
6. Informed consent from the patient or surrogate.
7. Patients can be treated within 90 minutes of the CT/CTA being completed.

Exclusion Criteria:

1. Hyperdensity on NCCT consistent with any intracranial hemorrhage. Any clinical suspicion of any intracranial hemorrhage even in the absence of visible blood on baseline brain imaging.
2. Large acute stroke >1/3 MCA territory or ASPECTS<5 visible on baseline CT scan.
3. Core of established infarction. No area of grey matter hypodensity at a similar or lesser density to white matter or in the judgment of the enrolling neurologist is consistent with a subacute ischemic stroke > 12 hours of age.
4. Clinical history, past imaging and clinical judgment suggest that the intracranial occlusion is chronic.
5. Patient is a candidate for and should receive standard of care IV tPA.
6. Stroke occurring as an in-patient. An in-patient is a person who has been officially admitted to the hospital to a ward bed. A patient in the ED who has not been formally admitted is still considered to be an outpatient.
7. Patient has a severe or fatal or disabling illness that will prevent improvement or follow-up or such that the treatment would not likely benefit the patient.
8. Patient cannot complete follow-up due to co-morbid non-fatal illness or is visiting the host sites city and cannot return for follow-up.
9. Pregnancy.
10. Patient is actively taking dual antiplatelet medication (aspirin & clopidogrel) in the last 48 hours.
11. International normalized ratio > 1.4
12. Standard thrombolysis exclusions (Taken from Canadian guidelines1)

NOTES: NIHSS = National Institutes of Health Stroke Scale ACA = anterior cerebral artery MCA = middle cerebral artery ICA = internal cerebral artery PCA = posterior cerebral artery VB = vertebrobasilar TICI = thrombolysis in cerebral ischemic scale CT = computed tomography NCCT = non-contrast CT CTA = CT angiography ASPECTS = Alberta Stroke Program Early CT Score IV = intravenous tPA = tissue plasminogen activator ED = Emergency Department

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Hill, MD,MSc FRCPC, Principal Investigator — University of Calgary; Shelagh B Coutts, MD,FRCPC, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Result] Coutts SB, Dubuc V, Mandzia J, Kenney C, Demchuk AM, Smith EE, Subramaniam S, Goyal M, Patil S, Menon BK, Barber PA, Dowlatshahi D, Field T, Asdaghi N, Camden MC, Hill MD; TEMPO-1 Investigators. Tenecteplase-tissue-type plasminogen activator evaluation for minor ischemic stroke with proven occlusion. Stroke. 2015 Mar;46(3):769-74. doi: 10.1161/STROKEAHA.114.008504. Epub 2015 Feb 12. PMID 25677596
- See also: TEMPO-1 site — http://www.ucalgary.ca/dcns/research/clinical_trials/TEMPO-1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from July 2012 through July 2014
Pre-assignment Details: All patients were treated with study drug.
Groups:
- Tenecteplase 0.1 mg/kg: 25 patients treated with 0.1 mg/kg intravenous tenecteplase
- Tenecteplase 0.25 mg/kg: 25 patients treated with 0.25 mg/kg intravenous tenecteplase
Period: Overall Study
Arm/Group | Tenecteplase 0.1 mg/kg | Tenecteplase 0.25 mg/kg
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Adults (age > 18) without an upper age limit, men and women with an acute ischemic stroke, less than 12 hours from symptom onset, who had a proven intracranial occlusion shown on CT angiography.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tenecteplase 0.1 mg/kg | Tenecteplase 0.25 mg/kg | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 15 | 16 | 31
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 72 [60 to 82] | 71 [61 to 81] | 71 [60 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 12 | 14 | 26
Region of Enrollment [Number; unit: participants]
  Canada | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Serious Bleeding Events
Description: The primary safety outcome will be the rate of expected serious adverse events associated with study drug. This will be defined as the number patients with at least one SAE divided by the number of patients enrolled by dose-tier. Thus, the unit of analysis will be the patient and not the SAE.
Time Frame: Up to 12 weeks
Population: All participants
Measure: Number; unit: Participants
Arm/Group | Tenecteplase 0.1 mg/kg | Tenecteplase 0.25 mg/kg
Number analyzed (Participants) | 25 | 25
Participants | 0 | 1

2. Secondary Outcome: Number of Patients With NIHSS 0 and mRS 0 and Barthel Index > 90
Description: Complete neurological and functional recovery at 90 days defined as: NIHSS 0 and mRS 0 iii)Complete neurological and functional recovery at 90 days defined as: a. NIHSS 0-1 and mRS 0-1 and Barthel Index > 90
  NIHSS = National Institutes of Health Stroke Scale. This integer scale ranges 0-42 and is a quantitative measure of the neurological examination.
  mRS = modified Rankin Scale. This integer scale ranges from 0-6 and is a criterion-based quantitative measure of functional neurological disability.
  BI = Barthel Index. This scale range from 0-100 (in increments of 5 points) and is a summative categorical score measuring activities of daily living.
Time Frame: 90 days
Population: All enrolled participants
Measure: Number; unit: Participants
Arm/Group | Tenecteplase 0.1 mg/kg | Tenecteplase 0.25 mg/kg
Number analyzed (Participants) | 25 | 25
Participants
  NIHSS = 0 at 90d | 15 | 19
  mRS = 0 at 90d | 10 | 14
  Barthel Index > 90 at 90d | 22 | 22

3. Other Pre Specified Outcome: Number of Patients With Recanalization 4-8 Hours Post-treatment
Description: Recanalization defined on follow-up 4-8 hour CTA as a modified arterial occlusive lesion (mAOL) score 0-1.
Time Frame: 4-8 hours
Population: 2 patients in each tier had missing data on this outcome.
Measure: Number; unit: Participants
Arm/Group | Tenecteplase 0.1 mg/kg | Tenecteplase 0.25 mg/kg
Number analyzed (Participants) | 23 | 23
Participants | 9 | 12

ADVERSE EVENTS:
Time Frame: 90 days from the date of enrolment
Description: Symptomatic intracranial hemorrhage
Arm/Group | Tenecteplase 0.1 mg/kg | Tenecteplase 0.25 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/25 | 1/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/25
Other Adverse Events (participants affected / at risk) | 12/25 | 8/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenecteplase 0.1 mg/kg (N=25) | Tenecteplase 0.25 mg/kg (N=25)
symptomatic intracerebral hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) — New posterior L temporal ICH (~15cc volume) with some associated sulcal SAH, contralateral to her stroke. New neurological deficits of aphasia. NIHSS remained at 4, but with different symptoms. Radiological classification rPH.
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenecteplase 0.1 mg/kg (N=25) | Tenecteplase 0.25 mg/kg (N=25)
Asymptomatic intracerebral hemorrhage (Nervous system disorders) | 1 (1) | 1
Atrial fibrillation (Cardiac disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 3 (3)
Carotid revascluarization (CEA or CAS) (Vascular disorders) | 2 (2) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 2 (2)
Bruising/hematoma (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
TEMPO-1 was a phase 2 study with a limited sample size. The program was designed to assess feasibility and safety and not efficacy. A further larger phase 3 study is planned.

Only selected adverse events are presented here. All SAEs are reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2012-06-06): https://cdn.clinicaltrials.gov/large-docs/45/NCT01654445/SAP_000.pdf